CLINICAL TRIAL: NCT07362719
Title: Therapeutic Efficacy of the Phlebology-oriented Thermal Cure at the Saint-Eloy Thermal Center in the Treatment of Symptoms of Severe Chronic Venous Insufficiency
Acronym: AMNEVILLE-PHL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société d'Exploitation des Thermes d'Amnéville (Other)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AMNEVILLE-PHL
Record Dates: First submitted 2026-01-13; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Venous Insufficiency of Leg
Keywords: Severe chronic venous insufficiency; Thermal cure; Phlebology; Balneology; Venous Insufficiency of Leg

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (with phlebology-oriented thermal cure) (Experimental): Participants suffering from severe chronic venous insufficiency receiving thermal treatment at the Saint-Eloy Thermal Center
  Interventions: Other: Phlebology oriented thermal cure
- Control (no thermal cure) (No Intervention): Participants suffering from severe chronic venous insufficiency without thermal treatment.

INTERVENTIONS:
Other: Phlebology oriented thermal cure — The phlebology oriented thermal cure takes place over a period of 3 consecutive weeks, with 6 days of cure per week (Monday to Saturday, i.e. 18 days). It includes 72 treatment sessions over the 18-day period and three medical consultations (including an initial consultation, a mid-course consultation, and a final consultation) organized by the resort's thermal doctors. The treatment program is established by the thermal doctor based on the patient's clinical profile.
  Arms: Interventional (with phlebology-oriented thermal cure)

SUMMARY:
Chronic venous insufficiency (CVI) is a common progressive vascular disease that affects nearly one-third of the French population. Despite considerable advances in the treatment of chronic venous insufficiency, this condition remains a burden for patients and national healthcare systems.

Balneotherapy-which includes thermal cures-is part of the therapeutic arsenal used in the treatment of chronic venous insufficiency. It is a relatively effective alternative with a relatively low cost compared to drug or surgical treatments. Phlebology is a thermal treatment orientation recognized by the French social security system.

The Saint-Eloy Thermal Center is listed among the thermal stations approved by the French Ministry of Health. It currently uses thermal water from Amnéville-les-Thermes to treat rheumatological and respiratory conditions, and wants to expand its range of orientations by adding phlebology. The AMNEVILLE-PHL study therefore aims to evaluate the efficacy and safety of the Saint-Eloy thermal cure for phlebology in patients suffering from severe chronic venous insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (≥ 18 years of age).
* Patients with severe chronic venous insufficiency of the lower limbs (C4a,b,c - C5 according to the CEAP (Clinical manifestations, Etiology, Anatomic distibution, Pathophysiology) classification (2020 revision) for at least one of the legs) confirmed by venous Doppler ultrasound of the lower limbs.
* Patients with an indication for a thermal cure exclusively focused on phlebology.
* Patients available to participate in a 3-week consecutive thermal cure at the Saint-Eloy Thermal Center, followed by 6 months of clinical follow-up, in accordance with the protocol schedule.
* Patients available to attend the visits scheduled in the protocol and able to complete the data collection documents.
* For women of childbearing age: patient using effective contraception.
* Patient affiliated with a health insurance plan or beneficiary (Art. L.1121-8-1, French Public Health Code).
* Patient who has given their informed consent in writing regarding their participation in the protocol.

Exclusion Criteria:

* Patients with a contraindication to thermal cure.
* Patients who have participated in thermal cure (regardless of type) within the last 9 months.
* Patients who have had an ulcer on their lower limbs that has healed within the last 3 months.
* Patients without venous trophic disorders of the lower limbs, and in particular patients with isolated class C3 chronic venous insufficiency or less in both lower limbs.
* Patients with an open ulcer on a lower limb (class C6).
* Patients for whom interventional venous treatment is due to begin within the next 6 months.
* Patients scheduled to undergo orthopedic surgery on the lower limbs within the next 6 months.
* Patients who are unable to walk.
* Patients with a known allergy to sulfur.
* Patients with any medically significant findings or significant history that may impact safety, interpretation of results, and/or subject participation in the study at 6 months, in the investigator's opinion.
* Patients simultaneously participating in another clinical trial or who have participated in another clinical trial for which the exclusion period has not ended.
* Vulnerable persons (Art. L.1121-5 to 8, and L1122-1-2, French Public Health Code).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy in relieving symptoms of severe chronic venous insufficiency | At baseline, at 3 months
  Measurement of the evolution in the modified Venous Clinical Severity Score (mVCSS ).
  The Venous Clinical Severity Score (VCSS) is composed of 10 items evaluating 8 clinical signs (pain, varicose veins, edema, skin pigmentation, inflammation, induration, ulcer, use of compression device). Each clinical sign is assessed on a scale of 0 to 3 (Absent (0), Mild (1), Moderate (2), Severe (3)) with a total VCSS score ranging from 0 to 30. The mVCSS excludes the item about the use of compression device because the thermal cure includes raising patient awareness about the importance of wearing compression devices. Thus, the modified VCSS score consists of 9 items with a total score ranging from 0 to 27. The lower the score, the fewer symptoms the patient has. The score is rated for both legs, but only the most severe leg based on the score at Baseline will be retained for the Primary Outcome Measure.
  The mVCSS is rated by an independant evaluator, and will be compared between both arms.

SECONDARY OUTCOMES:
Efficacy in relieving symptoms of severe chronic venous insufficiency | At baseline, at 3 months, at 6 months
  Measurement of the evolution in the mVCSS (modified Venous Clinical Severity Score), as described in the primary outcome measure.
  The modified VCSS score consists of 9 items with a total score ranging from 0 to 27. It is rated for both legs.
Efficacy in relieving symptoms of severe chronic venous insufficiency | At baseline, at 3 months, at 6 months
  Measurement of the evolution in the complete VCSS (Venous Clinical Severity Score).
  The complete VCSS is composed of 10 items evaluating 8 clinical signs (pain, varicose veins, edema, skin pigmentation, inflammation, induration, ulcer, use of compression device). Each clinical sign is assessed on a scale of 0 to 3 (Absent, Mild, Moderate, Severe) with a total VCSS score ranging from 0 to 30.
Pathology-related quality of life assessment | At baseline, at 3 months, at 6 months
  Self assessment of quality of life using the ChronIc Venous Insuficiency quality of life Questionnaire composed of 20 items (CIVIQ-20).
  The CIVIQ-20 is especially developped to assess the impact of chronic venous insufficiency on the patient's quality of life. A score will be calculated based on the questionnaire, from 20 to 100. The lower the score, the better the patient's quality of life.
Quality of life assessment | At baseline, at 3 months, at 6 months
  Self assessment of quality of life using the 5-dimension 5-level EuroQol (EQ-5D-5L) questionnaire, to assess the patient's general quality of life. The questionnaire consists of five questions (mobility, personal autonomy, daily activities, pain/discomfort, anxiety/depression) and a visual analog scale (VAS).
  For each patient, a health status (ranging from 11111 to 55555) will be obtained.
Impact on patient discomfort | At baseline, at 3 months, at 6 months
  Self assessment of the patient's discomfort intensity due to the chronic venous insufficiency, using a Visual Analog Scale (VAS) [10 cm line].
  A 10 cm line represents the intensity of the patient's discomfort. The patient places their discomfort on this line. 0 cm corresponds to a total absence of discomfort. 10 cm represents the worst discomfort the patient can imagine. The closer the patient places themselves to 10 cm, the worse their discomfort is.
Impact on skin pigmentation | At baseline, at 3 months, at 6 months
  Chromametric measurement on the calf skin using a chromameter.
Safety of Thermal Cure | Through study completion, an average of 6 months
  Adverse events and serious adverse events occurence. Skin, mobility, and vascular events are recorded.
Impact of the thermal cure focused on the the patient's clinical evolution assessed by the investigator | At 3 months, at 6 months
  Assessment of the clinical evolution by an independant evaluator using a 3-point Likert scale: better, neither better nor worse, worse.
Impact of the thermal cure focused on the the patient's clinical evolution self-assessed by the patient | At 3 months, at 6 months
  Self-assessment by the patient of his clinical evolution, using a 3-point Likert scale: better, neither better nor worse, worse.
Compliance for wearing compression devices | At baseline, at 3 months, at 6 months
  Assessment of the compliance for wearing compression devices using the "Compression therapy" item of the VCSS (Venous Clinical Severity Score), that goes from 0 to 3.
Patient satisfaction with the Saint-Eloy phlebology-oriented thermal cure | Between 3 weeks and 2 months
  Satisfaction questionnaire with 23 items for the patients of the interventionnal arm. The passation of the questionnaire is done at the end of the thermal cure.
  18 items use a numeric scale from 1 to 5 and 1 item use a numeric scale from 0 to 10. The minimal score is 18 and the maximal score is 100. The higher the score, the greater the patient satisfaction.
  2 items are binary closed questions (Yes/No). Positive responses correlate with patient satisfaction.
  2 items are optional open questions for positive or negative comments.
Medico-economic impact | At baseline, at 3 months, at 6 months
  Measurement of health care consumption and absenteeism at work through closed-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Claudine INVERNIZZI, Principal Investigator
Locations (1):
- Centre Thermal Saint-Eloy, Amnéville, France